CLINICAL TRIAL: NCT00851708
Title: Oxidative Stress and Postoperatory Renal Function in Deceased Kidney Transplantation
Brief Title: Impact of N-Acetylcysteine on Oxidative Stress and Renal Function in Deceased Kidney Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Antonio Marmo Lucon, University of São Paulo
Allocation: Randomized | Model: Parallel | Purpose: Prevention
Other Study IDs: NAC vs DKT; FAPESP 06/52046-0
Record Dates: First submitted 2009-02-25; First posted 2009-02-26 (Estimated); Last update posted 2009-03-02 (Estimated); Status verified 2009-02

CONDITIONS: Deceased Kidney Transplantation
Keywords: kidney; deceased kidney transplant; oxidative stress; renal function measurements
MeSH Terms: interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NAC (Active Comparator): treatment
  Interventions: Drug: N-acetylcysteine
- control (No Intervention)

INTERVENTIONS:
Drug: N-acetylcysteine — 600 mg bid orally from day 1 to 7 postoperative
  Arms: NAC

SUMMARY:
The aim of this interventional, prospective, randomized clinical trial is to evaluate the impact of the antioxidant N-acetylcysteine on oxidative stress in the first seven postoperative days and on renal function in the first three postoperative months in deceased kidney transplantation.

ELIGIBILITY:
Inclusion Criteria:

* First transplant
* Deceased kidney transplant

Exclusion Criteria:

* postoperative recovery at critical care unit
* illicit drug addiction
* psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Tiobarbituric acid reactive species measures | First seven postoperative days

SECONDARY OUTCOMES:
Serum creatinine | 7, 15, 30, 60, 90 postoperative day

CONTACTS AND LOCATIONS:
Locations (1):
- Clinics Hospital, University of Sao Paulo, Medical School, São Paulo, São Paulo, Brazil